CLINICAL TRIAL: NCT00095290
Title: Irbesartan Versus Placebo in Combination With Standard Cardiovascular Protection ACE-I Therapy With Ramipril for the Treatment of Albuminuria in Hypertensive Subjects at Elevated Cardiovascular Risk
Brief Title: Irbesartan Versus Placebo in Combination With Ramipril for Treatment of Albuminuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV131-169
Record Dates: First submitted 2004-11-02; First posted 2004-11-03 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2008-09

CONDITIONS: Albuminuria
Keywords: Albuminuria; Hypertension; Elevated Cardiovascular Risk; Albuminuria in Hypertensive Subjects at Elevated Cardiovascular Risk
MeSH Terms: conditions — Albuminuria; Hypertension | interventions — Ramipril; Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: Ramipril + Irbesartan
- A2 (Placebo Comparator)
  Interventions: Drug: Ramipril + Placebo

INTERVENTIONS:
Drug: Ramipril + Irbesartan — Tablets + Capsules, Oral, 10mg Ramipril + 300mg Irbesartan target dose, Once daily, 20 weeks.
  Other Names: Avapro
  Arms: A1
Drug: Ramipril + Placebo — Tablets + Capsules, Oral, 10mg Ramipril + 300mg Placebo target dose, Once daily, 20 weeks.
  Arms: A2

SUMMARY:
Albumin in the urine is usually a signal that you might be at risk of cardiovascular complications. The purpose of this study is to determine if the albumin in your urine can be decreased by the treatment regimen that consists of irbesartan taken at the same time with ramipril.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to provide written informed consent.
* Males and Females 55 years of age and over
* Subjects must have a history of high blood pressure and elevated cardiovascular risk defined as one of the following:

  1. Diabetes
  2. Advanced coronary disease defined as previous myocardial infarction. Active angina, or significant changes in tests indicating ischemia
  3. Artery disease in the legs, limiting walking capacity and/or blood flow in the legs
  4. Stroke occurring more than 3 months prior to the screening visit
* All subjects must also have albuminuria (protein in the urine) that is confirmed by a urine test at the first study visit.
* All subjects must currently be treated with a class of drugs called ACE inhibitors (e.g., benazepril, captopril, enalapril, lisinopril, moexipril, ramipril, quinapril, perindopril) for at least 2 months prior to the study.
* Women of childbearing potential (WOCBP) must be using adequate methods of contraception to avoid pregnancy throughout the study and four weeks after the study ends.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Acute systemic febrile/infectious disease or infectious or inflammatory disease of the kidneys
* Narrowing of the kidney arteries
* Hypotension (low blood pressure) or very high blood pressure
* Moderate or Severe Heart Failure
* Chronic autoimmune disease
* Cancer unless cured or no further treatment needed
* Severe kidney failure
* Allergy to drugs used in the study: ARBs (candesartan, irbesartan, losartan, telmisartan, valsartan, and/or any other ARB currently or previously in development) and ACE-inhibitors (benazepril, captopril, enalapril, lisinopril, moexipril, ramipril, quinapril, perindopril)
* Administration of any other investigational drug within 30 days of planned enrollment into the study.
* Any circumstances that would prevent coming for study visits or taking study drugs

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change in AER from baseline to Week 20

SECONDARY OUTCOMES:
Change from baseline in seated systolic and diastolic blood pressures at Week 20; Comparison of change from baseline in seated systolic and diastolic blood pressures at Week 20 between treatment groups

CONTACTS AND LOCATIONS:
Locations (92):
- United States (11):
  - Local Institution, Tustin, California
  - Local Institution, Miami, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Flushing, New York
  - Local Institution, New York, New York
  - Local Institution, Cleveland, Ohio
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, San Antonio, Texas
  - Local Institution, Milwaukee, Wisconsin
- Australia (9):
  - Local Institution, Burwood, New South Wales
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Gosford, New South Wales
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Box Hill, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Parkville, Victoria
  - Local Institution, Fremantle, Western Australia
- Canada (8):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Scarborough Village, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Laval, Quebec
  - Local Institution, Longueuil, Quebec
- France (5):
  - Local Institution, Boulogne-sur-Mer
  - Local Institution, Colmar
  - Local Institution, Grenoble
  - Local Institution, Pessac
  - Local Institution, Strasbourg
- Germany (9):
  - Local Institution, Aschaffenburg
  - Local Institution, Bad Mergentheim
  - Local Institution, Göttingen
  - Local Institution, Halle
  - Local Institution, Künzing
  - Local Institution, München
  - Local Institution, Ornbau
  - Local Institution, Vellmar
  - Local Institution, Villingen-Schwenningen
- Israel (12):
  - Local Institution, Ashkelon
  - Local Institution, Beersheba
  - Local Institution, Hadera
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Kiryat Biyalik
  - Local Institution, Nazareth
  - Local Institution, Ramat Gan
  - Local Institution, Rehovot
  - Local Institution, Tel Aviv
  - Local Institution, Ẕerifin
- Italy (7):
  - Local Institution, Chieri
  - Local Institution, Genova
  - Local Institution, Lecco
  - Local Institution, Napoli
  - Local Institution, Rimini
  - Local Institution, Rome
  - Local Institution, San Benedetto del Tronto
- Latvia (2):
  - Local Institution, Daugavpils
  - Local Institution, Riga
- Lithuania (5):
  - Local Institution, Kaunas
  - Local Institution, Klaipėda
  - Local Institution, Panevezys
  - Local Institution, Šiauliai
  - Local Institution, Vilnius
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, México, San Lis Potosi
- Netherlands (7):
  - Local Institution, Amsterdam
  - Local Institution, Blaricum
  - Local Institution, Eindhoven
  - Local Institution, Groningen
  - Local Institution, Stadskanaal
  - Local Institution, Zeist
  - Local Institution, Zwolle
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Spain (5):
  - Local Institution, Barcelona
  - Local Institution, Jerez de la Frontera
  - Local Institution, Las Palmas de G. C.
  - Local Institution, Madrid
  - Local Institution, Marbella
- United Kingdom (4):
  - Local Institution, Middlesbrough, Cleveland
  - Local Institution, Belfast, County Durham
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Derby, West Midlands

REFERENCES:
- [Derived] Bakris GL, Ruilope L, Locatelli F, Ptaszynska A, Pieske B, de Champlain J, Weber MA, Raz I. Treatment of microalbuminuria in hypertensive subjects with elevated cardiovascular risk: results of the IMPROVE trial. Kidney Int. 2007 Oct;72(7):879-85. doi: 10.1038/sj.ki.5002455. Epub 2007 Aug 1. PMID 17667984